CLINICAL TRIAL: NCT02479009
Title: Fluoroscopy vs. Computed Tomography for Diagnosis of Displacement and Instability of Acute Scaphoid Waist Fractures
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The investigator left the institution so the study was terminated.
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Skane University Hospital (Other); Ghaem Hospital (Other)
Responsible Party: Principal Investigator, David C. Ring, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014P002038
Record Dates: First submitted 2015-06-19; First posted 2015-06-23 (Estimated); Last update posted 2016-12-22 (Estimated); Status verified 2016-12

CONDITIONS: Acute Scaphoid Waist Fractures
MeSH Terms: interventions — Fluoroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Fluoroscopy — Each patient will undergo fluoroscopy-imaging evaluation in the office to determine whether the fracture moves (instability). The investigators will deviate the wrist from ulnar to radial and back in posteroanterior, oblique and lateral views with the wrist in neutral flexion. Any angulation or translation at the fracture site or more than one millimeter displacement or gap will be considered as a sign of instability. The fluoroscopy will be viewed and an image showing the largest gap will be saved. The diagnosis of instability (which is the same as displacement with this test) will be made by consensus of the research team.

SUMMARY:
Aim:

The aim of this study is to analyze if fluoroscopy is as accurate as computed tomography in diagnosing displacement of acute scaphoid waist fractures.

Primary null hypothesis:

Fluoroscopy has comparable sensitivity, specificity, accuracy, positive and negative predictive values compared with computed tomography for the diagnosis of displacement of acute scaphoid waist fractures.

Secondary null hypothesis:

All fractures diagnosed as non-displaced and treated without surgery are healed on radiographs and discharged from care within 6 months of injury.

DETAILED DESCRIPTION:
The only confirmed risk factor for nonunion of a scaphoid waist fracture is displacement. There is consensus that displaced fractures should be treated with open or arthroscopically assisted reduction and internal fixation (ORIF). However, the optimal method to diagnose displacement is debated. Radiographic, computed tomography (CT), and arthroscopic diagnostic criteria for the diagnosis of displacement exist. There is no consensus regarding the imaging modality and measurements to use to diagnose scaphoid displacement. The definition of displacement in recent randomized trials is incompletely described and inconsistent. Fluoroscopy is more convenient, less expensive, and uses less radiation than CT scanning. If displaced fractures are unstable, then this should be apparent on fluoroscopy. The aim of this study is to analyze if fluoroscopy is as accurate as computed tomography in diagnosing displacement of acute scaphoid waist fractures.

ELIGIBILITY:
Inclusion Criteria:

* All patients (>18 years) with a radiographically visible acute (< 2 weeks since injury) scaphoid waist fracture will be included. The subject has to speak and write English or Spanish fluently to be able to provide informed consent

Exclusion Criteria:

* Pregnant women
* Women who are capable of becoming pregnant and not on birth control will be excluded due to the risk of pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-06; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Accuracy of Fluoroscopy | Less than 2 weeks from injury date
  The reference standard for calculation of diagnostic performance characteristics of fluoroscopy will be displacement on CT scanning defined as follows: Displacement on CT scan defined as any angulation or translation, or greater than 1mm gap at any point in the fracture line.

CONTACTS AND LOCATIONS:
Overall Officials: David Ring, MD, PhD, Principal Investigator — Massachusetts General Hospital